CLINICAL TRIAL: NCT02147522
Title: A Helping Hand (AHH) to Activate Patient-Centered Depression Care Among Low-Income Patients
Brief Title: A Helping Hand Among Low-Income Patients
Acronym: AHH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Kathleen R. Ell, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AD-1304-7364
Record Dates: First submitted 2014-05-19; First posted 2014-05-26 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-04

CONDITIONS: Depression; Diabetes; Heart Disease
Keywords: community health worker; promotoras; self-care behaviors activation; depression; low-income patients; safety-net care
MeSH Terms: conditions — Depression; Diabetes Mellitus; Heart Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A Helping Hand (AHH) (Experimental): Participants receive DHS-PCMH usual care from their respective county health clinic providers plus the AHH intervention provided by study promotoras. AHH intervention includes 6 weekly in-person or via-telephone intervention sessions followed by 3 monthly telephone booster sessions aimed at reducing the burden and strain on patients, families, and care providers by assessing, enhancing, and facilitating patient depression and co-morbid illness self-care management, and activating patient communication with clinic medical providers.
  Interventions: Behavioral: Self-care management
- Usual Care (UC) (No Intervention): Participants receive DHS Patient Centered Medical Home (PCMH) clinic team usual care from their respective county health clinic providers.
  PCMH model has available DHS medical providers and social workers for depression care and refer patients when indicated to community mental health clinics. Problem-Solving Therapy (PST) is available in some of participating clinics.

INTERVENTIONS:
Behavioral: Self-care management — AHH behavioral intervention is provided by promotoras
  Arms: A Helping Hand (AHH)

SUMMARY:
Study Hypotheses (Ho) and Research Questions (RQ):

* Ho1. AHH will significantly improve patient depression treatment acceptance/adherence and depression symptoms vs UC at 6 and 12 months post-baseline.
* Ho2. A Helping Hand (AHH) will significantly improve and sustain patient self-care management in Self-Efficacy for Managing Chronic Disease (SEMCD) and Quality of Life vs UC at 6 and 12 months post-baseline.
* RQ1. What is the association between depression symptoms and concurrent chronic illness self-care management over time by group?
* RQ2. Will AHH reduce hospitalizations and Emergency Room visits and improve clinic appointment-keeping?
* RQ3. Will patient care satisfaction and reported barriers to self-care management vary by study group?
* RQ4. What factors are identified via qualitative assessments of patients, promotoras, Department of Health Services (DHS) medical and social work providers, and DHS clinic/organizational leadership regarding satisfaction with, sustainable uptake of, and suggested modifications of the AHH promotora delivery model?
* RQ5. What potential technology applications would enhance promotoras delivering patient-centered self-care training and resource navigation, communicating and integrating care with DHS, and disseminating AHH?

DETAILED DESCRIPTION:
Major depression, plus other chronic illness such as diabetes, coronary heart disease and heart failure is common among low-income, culturally diverse safety net care patients. Unfortunately, many of these patients are uncomfortable about either asking their doctor questions about their illness and treatment options and their illness self-care or informing their doctors about their treatment preferences. Lack of strong engagement with medical providers occurs because patients believe they lack the knowledge to ask questions or to understand and follow recommended self-care and their concern that their medical provider lacks understanding of their treatment preferences. These factors often result in patient worry, poor adherence to prescribed treatment, and worsening illness status and even early death. The study will be conducted by a university, the Los Angeles County Department of Health Services (DHS) and a community health worker organization research team. The study will be conducted within two DHS Patient-Centered Medical Home clinics, with each patient having a designated primary care team of physician, nurse, social worker and medical assistant. Study patients with major depression and other illnesses face numerous self-care management barriers: managing concurrent symptoms (depression, pain, anxiety etc.) and cultural influences (depression stigma, diet), difficulty in navigating primary and specialty doctor and treatment plans, while at the same time experiencing daily social and economic stress. The randomized comparative effectiveness study plans to recruit 350 patients with major depression and a concurrent chronic illness (i.e., diabetes, heart failure, coronary heart disease) from two DHS PCMH community health centers. To enhance patient-centered research community partnerships, patients will be provided A Helping Hand (AHH) in which a community organization- based promotora aims to activate patient-centered depression self-care training and practical assistance to: a) improve and personalize major depression self-care (e.g., medication or psychotherapy preference, treatment adherence, fatigue, pain, diet, activity, stress management, family/caregiver communication); b) activate patient-provider communication, clinic appointment keeping and treatment coordination; and c) and facilitate patient navigation and receipt of needed community resources. AHH aims to improve patient self-care management and patient-provider care management relationships among underserved low-income patients, who must simultaneously cope with major depression and chronic co-morbid physical illness. Study objectives aim to determine: 1) whether community health worker promotora care management training improves patient-centered outcomes, such as self-care need and management, treatment adherence, symptom improvement, and care satisfaction over the usual team care; 2) depression symptom improvement; and 3) patient hospitalizations and ER visits frequency.

ELIGIBILITY:
Inclusion Criteria:

* age >=18 years, have a phone, meet PHQ-9 score of 10 or more, and have concurrent diabetes, CHD, or HF.

Exclusion Criteria:

* current suicidal ideation,inability to speak either English or Spanish fluently, a score of 2 or greater on the CAGE 4M alcohol assessment,recent use of lithium or antipsychotic medication, and cognitive impairment precluding informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2013-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Ell, DSW, Principal Investigator — USC Suzanne Dworak-Peck School of Social Work
Locations (3):
- United States (3):
  - El Monte Comprehensive Health Center, El Monte, California
  - H. Claude Hudson Comprehensive Health Center, Los Angeles, California
  - Edward R. Roybal Comprehensive Health Center, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh H, Ell K. Associations Between Changes in Depressive Symptoms and Social Support and Diabetes Management Among Low-Income, Predominantly Hispanic Patients in Patient-Centered Care. Diabetes Care. 2018 Jun;41(6):1149-1156. doi: 10.2337/dc17-2000. Epub 2018 Mar 27. PMID 29588293
- [Derived] Ell K, Aranda MP, Wu S, Oh H, Lee PJ, Guterman J. Promotora assisted depression and self-care management among predominantly Latinos with concurrent chronic illness: Safety net care system clinical trial results. Contemp Clin Trials. 2017 Oct;61:1-9. doi: 10.1016/j.cct.2017.07.001. Epub 2017 Jul 3. PMID 28684357
- [Derived] Ell K, Aranda MP, Wu S, Oh H, Lee PJ, Guterman J. Promotora assisted depression care among predominately Hispanic patients with concurrent chronic illness: Public care system clinical trial design. Contemp Clin Trials. 2016 Jan;46:39-47. doi: 10.1016/j.cct.2015.11.012. Epub 2015 Nov 17. PMID 26600285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were identified from medical charts or referred by care providers at three LAC-DHS community clinics with Patient Centered Medical Home (PCMH) care model, screened and recruited between April 2014 to May 2015.
Groups:
- A Helping Hand (AHH): Participants received PCMH depression care services from their respective county health clinic providers plus the AHH intervention. Promotoras provided 6 weekly in-person or via-telephone intervention followed by 3 monthly telephone sessions aimed at reducing the burden and strain on patients, families, and care providers by assessing, enhancing, and facilitating patient depression and co-morbid illness self-care management, and activating patient communication with clinic medical providers.
- Usual Care (UC): Participants received DHS Patient Centered Medical Home (PCMH) clinic usual care from their respective county health clinic providers.
  PCMH model has available DHS medical providers and social workers for depression care and refer patients when indicated to community mental health clinics. Problem-Solving Therapy (PST) is available in some of participating clinics.
Period: Overall Study
Arm/Group | A Helping Hand (AHH) | Usual Care (UC)
Started | 178 | 170
Completed | 122 | 122
Not Completed | 56 | 48

BASELINE CHARACTERISTICS:
Population: From April 2014 to May 2015, 1957 were screened, 22% met criteria for major depression. Of 421 study eligible, 354 patients agreed to participate but 6 did not complete the baseline assessment. It yielded a final valid enrollment number N=348, with178 (51%) randomized to the AHH intervention group and 170 (49%) to the comparison UC group.
Groups:
- A Helping Hand (AHH): Participants received DHS-PCMH usual care from their respective county health clinic providers plus the AHH intervention provided by study promotoras. AHH intervention includes 6 weekly in-person or via-telephone intervention sessions followed by 3 monthly telephone booster sessions aimed at reducing the burden and strain on patients, families, and care providers by assessing, enhancing, and facilitating patient depression and co-morbid illness self-care management, and activating patient communication with clinic medical providers.
- Usual Care (UC): Participants received DHS Patient Centered Medical Home (PCMH) clinic team usual care from their respective county health clinic providers.
  PCMH model has available DHS medical providers and social workers for depression care and refer patients when indicated to community mental health clinics. Problem-Solving Therapy (PST) is available in some of participating clinics.
- Total: Total of all reporting groups
Arm/Group | A Helping Hand (AHH) | Usual Care (UC) | Total
Number analyzed (Participants) | 178 | 170 | 348
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.77 (8.79) | 56.31 (8.47) | 56.54 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 144 | 296
  Male | 26 | 26 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 176 | 168 | 344
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 178 | 170 | 348
Depression Severity, Categorial [Count of Participants; unit: Participants]
  Moderate, PHQ-9 score 10-14 | 71 | 62 | 133
  Moderately severe, PHQ-9 score 15-19 | 74 | 73 | 147
  Severe, PHQ-9 score 20+ | 33 | 35 | 68

OUTCOME MEASURES:

1. Primary Outcome: Response Rate - 50 Percent or Greater Reduction in Patient Health Survey-9 (PHQ-9) Score Since Baseline
Description: The PHQ-9, which establishes provisional depressive disorder diagnosis as well as grades depressive symptom severity, will be obtained from all study subjects at recruitment and during the four waves of data collection (up to 12 months). The PHQ-9 scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day), with possible scores ranging from 0 to 27, with cut points of 5,10,15, and 20 representing the thresholds for mild, moderate, moderately severe, and severe depression. A validated Spanish version of the PHQ-9 will be used. Clinically meaningful improvement of depressive symptoms was assessed as a ≥50% score reduction since baseline assessment.
Time Frame: 6- and12-month follow-ups
Population: Analyses for hypothesis testing related to the evaluation of AHH effects were carried out according to the intention-to-treat rule consistent with standard practice in clinical trials.
Measure: Count of Participants; unit: Participants
Arm/Group | A Helping Hand (AHH) | Usual Care (UC)
Number analyzed (Participants) | 130 | 133
Participants
  6-Month | 69 | 68
  12-Month: number analyzed (Participants) | 122 | 122
  12-Month | 67 | 60

2. Secondary Outcome: Change From Baseline in MOS Short-Form Health Survey Physical Component Summary (PCS)
Description: The Physical Component Summary (PCS) is a norm-based score standardized to the general U.S. population with a mean of 50, and a SD of 10. Scores range from 0 to 100, a higher score indicating better physical health.
Time Frame: baseline, 6- and 12-month follow-ups
Population: Some participants did not complete follow-up assessments (6-month: 48 AHH and 37 UC; 12-month: 56 AHH and 48 UC).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Helping Hand (AHH) | Usual Care (UC)
Number analyzed (Participants) | 178 | 170
units on a scale
  Baseline | 38.28 (10.45) | 38.27 (11.14)
  6-Month: number analyzed (Participants) | 130 | 133
  6-Month | 37.85 (11.2) | 36.33 (11.35)
  12-Month: number analyzed (Participants) | 122 | 122
  12-Month | 37.63 (10.73) | 37.1 (11.68)

3. Other Pre Specified Outcome: Change From Baseline in Self-Efficacy for Managing Chronic Disease (SEMCD) Score
Description: The Self-Efficacy for Managing Chronic Disease (SEMCD) contains 6 items that are common across chronic diseases: symptom control, role function, emotional functioning and communicating with physicians, rated in a scale 1 (not at all confident) to 10 (totally confident). The score for the scale is the mean of the six items. Higher number indicates higher self-efficacy.
Time Frame: baseline, 6- and 12-month follow-ups
Population: Some participants did not complete follow-up assessments (6-month: 48 AHH and 37 UC; 12-month: 56 AHH and 48 UC).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A Helping Hand (AHH) | Usual Care (UC)
Number analyzed (Participants) | 178 | 170
units on a scale
  Baseline | 6.22 (3.1) | 5.8 (2.62)
  6-Month: number analyzed (Participants) | 130 | 133
  6-Month | 7.2 (2.73) | 6.85 (2.89)
  12-Month: number analyzed (Participants) | 122 | 122
  12-Month | 7.23 (2.68) | 6.79 (3.0)

ADVERSE EVENTS:
Time Frame: 1 year
Description: The study intervention provided only educational sessions, thus no serious and other non-serious adverse events were collected or assessed systematically. However, we documented event information revealed by family member of participants, if any.
Arm/Group | A Helping Hand (AHH) | Usual Care (UC)
All-Cause Mortality (participants affected / at risk) | 0/178 | 1/170
Serious Adverse Events (participants affected / at risk) | 2/178 | 2/170
Other Adverse Events (participants affected / at risk) | 0/178 | 0/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A Helping Hand (AHH) (N=178) | Usual Care (UC) (N=170)
Death (General disorders) | 0 (0) | 1 (1) — revealed by family member who did not specify the cause
Hospitalization (General disorders) | 1 (1) | 1 (1)
Resided in a nursing home (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
1) patients lost follow up in intervention visits, outcome interviews; 2) community health workers activated in DHS-PCMH at the same time the AHH trial started; 3) reliance on self-reported outcomes while DHS medical records system update was delayed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No